CLINICAL TRIAL: NCT04347538
Title: Impact of Nasal Saline Irrigations on Viral Load in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Justin Turner, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200693
Record Dates: First submitted 2020-04-11; First posted 2020-04-15 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients enrolled will be randomized to one of three treatment groups (1. control- no intervention, 2. intervention 1 - nasal saline irrigations BID, 3. intervention 2- nasal saline irrigations with ½ teaspoon surfactant (Johnson's baby shampoo) BID).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group, No intervention (No Intervention): control group, no nasal irrigation
- Saline Nasal Irrigation (Experimental): Nasal irrigation BID with normal saline
  Interventions: Other: Saline Nasal Irrigation
- Saline with Baby Shampoo Nasal Irrigation (Experimental): Nasal irrigation BID with normal saline and 1/2 teaspoon baby shampoo
  Interventions: Other: Saline with Baby Shampoo Nasal Irrigation

INTERVENTIONS:
Other: Saline Nasal Irrigation — Saline nasal irrigation BID
  Arms: Saline Nasal Irrigation
Other: Saline with Baby Shampoo Nasal Irrigation — Saline with 1/2 teaspoon Baby Shampoo Nasal Irrigation.
  Arms: Saline with Baby Shampoo Nasal Irrigation

SUMMARY:
Nasal saline irrigations are a safe and commonly used mechanism to treat a variety of sinonasal diseases including sinusitis, rhinitis, and upper respiratory tract infections. When used properly, these irrigations are a safe and easy intervention available over the counter without a prescription. Additionally, baby shampoo has been found to be a safe additive functioning as a surfactant when a small amount is added to the saline rinses which may help augment clearance of the sinonasal cavity.

While many systemic medications and treatments have been proposed for COVID-19, there has not yet been a study looking at targeted local intervention to the nasal cavity and nasopharynx where the viral load is the highest. Studies have shown that the use of simple over the counter nasal saline irrigations can decrease viral shedding in the setting of viral URIs, including the common coronavirus (not SARS-CoV-2). Further, as SARS-CoV-2 is an enveloped virus, mild-detergent application with nasal saline would neutralize the virus further. It is our hypothesis that nasal saline or nasal saline with baby shampoo irrigations may decrease viral shedding/viral load and viral transmission, secondary bacterial load, nasopharyngeal inflammation in patients infected with the novel SARS-CoV-2.

DETAILED DESCRIPTION:
The novel coronavirus known as SARS-CoV-2 and the associated disease process COVID-19 (coronavirus disease 2019) was first seen in late 2019 in Wuhan, China. Over the following months, it quickly spread across the continent and, in short order, the globe, making an impact that hasn't been seen in generations. Although coronaviruses have been prevalent for millennia, this version is immunologically novel, and thus there is no natural immunity to the virus. This has been a major reason for its rapid spread across the world.

Previous members of the coronavirus family have typically caused upper respiratory symptoms such as the common cold, though there have also been more virulent versions of this virus seen in the recent past, such as SARS (Severe Acute Respiratory Syndrome) and MERS (Middle East Respiratory Syndrome). Similarly named, SARS-CoV-2 also causes upper respiratory symptoms but has varied from the previous viral syndromes in a number of ways including how quickly it has been able to transmit within a population. This is a disease that does not segregate and can affect all ages, genders, and ethnicities. Everyone is susceptible to this virus.

New diagnostic and therapeutic approaches for respiratory viruses are also being rapidly developed and polymerase chain reaction-based (PCR) diagnostics and multiplex assays are increasingly used in clinical laboratories for SARS-CoV-2 clinical detection and subtyping. Rapid antigenic and genetic evolution has been expected for SARS-CoV-2 strains, and a better understanding of SARS-CoV-2 evolutionary dynamics is needed to establish an effective vaccine.

Our present understanding of the nature and extent of the upper respiratory track (URT) microbiome in humans is limited. Furthermore, we have little understanding of how acute viral respiratory infections of SARS-CoV-2 influence the URT microbiome, or how genotypic differences in the virus influence the URT microbiome and vice versa. Innate immune responses to pathogens, along with dysregulation of inflammation, are key factors involved in pathogenesis, and different viral pathogens activate different types of inflammatory responses. Respiratory viral infection i.e., SARS-CoV-2 infection is expected to activate TLR2, TLR3, TLR4 and TLR7 responses and this is likely to modulate commensal microbiota populations. It is not yet known if the severity of SARS-CoV-2 disease in older adults is due to a biased host response, SARS-CoV-2 virulence determinants, or the impact infection has on commensal microbiota.

Up to this point, there is no unanimously approved treatment for the disease nor is there a vaccine or antiviral drugs available for the public. The primary methods for treatment of this deadly virus have been supportive in nature including intubation in severe cases with respiratory failure.

While a unanimous treatment has yet to be discovered, there has been a great amount of knowledge garnered over the last few months about the virus and the disease that accompanies it. Several studies have demonstrated high viral titers within the nasopharynx and oral cavity and many have posited that this is the primary source of infection and viral replication. Additionally, a high nasal/nasopharyngeal viral load has been associated with increased symptoms and higher severity of the disease.

Interestingly, there have been a number of studies recently looking at the effect of nasal saline irrigations in the setting of viral URIs, including coronaviruses (not including SARS-CoV-2). One of the major takeaways from these studies was decreased viral shedding in patients treated with saline irrigations compared to the control group. Nasal saline irrigations are available over the counter and widely viewed as both safe and affordable. Could these irrigations have a similar effect on the novel SARS-CoV-2 that they have on other viral respiratory infections?

ELIGIBILITY:
Inclusion Criteria:

* Patients testing positive for COVID-19 at Vanderbilt University Medical Center or VUMC-associated testing centers
* Age of 18 years or greater
* Patients must be planning self-quarantine after infection in the greater Nashville area within a 30-mile radius of Vanderbilt University Medical Center

Exclusion Criteria:

* Requiring hospitalization - only outpatient COVID-19 cases are eligible for the study
* Current use of nasal saline irrigations or other intranasal medications
* Inability to perform saline irrigations/nasal swabs in separate bathroom away from household contacts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kimura, MD, Principal Investigator — Vanderbilt University Medical Center; Justin H. Turner, MD, PhD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderblt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esther CR Jr, Kimura KS, Mikami Y, Edwards CE, Das SR, Freeman MH, Strickland BA, Brown HM, Wessinger BC, Gupta VC, Von Wahlde K, Sheng Q, Huang LC, Bacon DR, Kimple AJ, Ceppe AS, Kato T, Pickles RJ, Randell SH, Baric RS, Turner JH, Boucher RC. Pharmacokinetic-based failure of a detergent virucidal for severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) nasal infections: A preclinical study and randomized controlled trial. Int Forum Allergy Rhinol. 2022 Sep;12(9):1137-1147. doi: 10.1002/alr.22975. Epub 2022 Jan 31. PMID 35040594

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline With Baby Shampoo Nasal Irrigation | Saline Nasal Irrigation | Control Group, No Intervention
Started | 28 | 29 | 31
Completed | 24 | 24 | 24
Not Completed | 4 | 5 | 7
Not completed — Lost to Follow-up | 4 | 5 | 7

BASELINE CHARACTERISTICS:
Population: Baseline data is available only for those who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline With Baby Shampoo Nasal Irrigation | Saline Nasal Irrigation | Control Group, No Intervention | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 23 | 70
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (18) | 39 (15) | 39 (15) | 39 (23)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis population includes those who were screened, enrolled, and completed follow up. Data on participant sex was only collected for 72 participants.
  Participants
    Female | 15 | 12 | 10 | 37
    Male | 9 | 12 | 14 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Viral Load in the Nasopharynx Over the Course of COVID-19 Infection
Description: Perform qPCR Analysis to asses viral shedding over 21 day study period. Data expressed as viral shedding of N1 protein. Viral shedding = log10(change values at first day to the max value of Ct)/days between two values.
Time Frame: Day 1 to day 21
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL/days
Arm/Group | Saline With Baby Shampoo Nasal Irrigation | Saline Nasal Irrigation | Control Group, No Intervention
Number analyzed (Participants) | 24 | 24 | 24
Log10 copies/mL/days | .116 [-.031 to 0.333] | .071 [-.047 to .253] | .118 [-.083 to .330]

2. Secondary Outcome: Symptom Assessment Via Wisconsin Upper Respiratory System Survey 21 With Additional Symptoms Prevalent During SARS-CoV-2
Description: Identify symptom burden at day 5 using the modified Wisconsin Upper Respiratory System Survey 21. Minimum = 0. Maximum =21. Higher scores represent a worse outcomes.
Time Frame: 21 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline With Baby Shampoo Nasal Irrigation | Saline Nasal Irrigation | Control Group, No Intervention
Number analyzed (Participants) | 24 | 24 | 24
score on a scale | 13 (14) | 16.3 (17.8) | 16.4 (11.8)

ADVERSE EVENTS:
Time Frame: Adverse events collected from time of consent through study completion, approximately 21 days after enrollment.
Description: Adverse events reports to be to the Vanderbilt HRPP as required per institutional policy.
Arm/Group | Control Group, No Intervention | Saline Nasal Irrigation | Saline With Baby Shampoo Nasal Irrigation
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT04347538/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04347538/ICF_000.pdf